CLINICAL TRIAL: NCT03880045
Title: Topical Tranexamic Acid Plus Perivascular Vasopressin to Decrease Bleeding at the Time of Abdominal Myomectomy: A Double-blinded Randomized Placebo-controlled Trial
Brief Title: Topical Tranexamic Acid Plus Perivascular Vasopressin at the Time of Abdominal Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/206/19
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Myoma
Keywords: abdominal myomectomy; tranexamic acid; vasopressin
MeSH Terms: conditions — Myoma; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: A double-blinded randomized controlled stud
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blinded randomized controlled stud
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical TA plus vasopressin (Active Comparator): Intraoperative perivascular injection of one ampoule of vasopressin containing 20 units in 1 ml after dilution in 19 ml of normal saline during myomectomy plus gauze soaked with 2 g tranexamic acid (20 ml) diluted in 100 ml of sodium chloride0.9%
  Interventions: Drug: Topical TA; Drug: vasopressin
- placebo to TA plus vasopressin (Active Comparator): Intraoperative perivascular injection of one ampoule of vasopressin containing 20 units in 1 ml after dilution in 19 ml of normal saline during myomectomy plus placebo to tranexamic acid
  Interventions: Drug: vasopressin; Other: placebo to TA

INTERVENTIONS:
Drug: Topical TA — A gauze soaked with 2 g tranexamic acid (20 ml) diluted in 100 ml of sodium chloride0.9%
  Other Names: Active comparator
  Arms: Topical TA plus vasopressin
Drug: vasopressin — intraoperative perivascular injection of one ampoule of vasopressin containing 20 units in 1 ml after dilution in 19 ml of normal saline during myomectomy
  Other Names: Active Comparator
Other: placebo to TA — (120 ml of sodium chloride 0.9%) used to compress the myoma bed for 5 min.
  Other Names: placebo comparator
  Arms: placebo to TA plus vasopressin

SUMMARY:
In this study, the investigators will investigate the effectiveness of a topical tranexamic acid plus perivascular vasopressin compared with perivascular vasopressin alone for the reduction of blood loss at the time of myomectomy

DETAILED DESCRIPTION:
Uterine fibroids are the most common female pelvic tumors occurring in about 15% to 30% of women in the reproductive age group. The major problem with myomectomy is excessive bleeding from the increased uterine blood supply. This can be life-threatening, resulting in blood transfusions, febrile morbidity, and potentially in loss of reproductive potential from a hysterectomy. Knowledge of the effectiveness of the interventions used to reduce blood loss during myomectomy is essential to enable evidence-based clinical decisions. Topical application of tranexamic acid(TA) provides a high drug concentration at the site of the wound and a low systemic concentration. Studies from cardiac and orthopedic surgery have shown an equal or superior effect of topical compared with intravenous TA on both bleeding and transfusion requirement. Topical treatment is cost-effective, and adverse effects or drug interactions have not been reported

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for abdominal myomectomy with documented uterine fibroids on pelvic imaging
* Age ≥ 18 years and ≤ 50 years
* Pre-operative hemoglobin >8 g/dl
* Ability to understand and the willingness to sign a written informed consent.
* Admissible medical/surgical history
* Five or less symptomatic uterine myomas
* All myomas are subserous or intramural.
* Uterine size less than 24 weeks of pregnancy

Exclusion Criteria:

* Patients who have had a prior abdominal myomectomy
* Post-menopausal women
* Patients with known bleeding/clotting disorders
* Patients with a history of gynecologic malignancy
* Hypertension.
* Cardiac and Pulmonary Diseases.
* Obesity (body mass index > 30 kg/m2).
* History of allergic reactions attributed to misoprostol
* Cases that will require intraoperative conversion of myomectomy to hysterectomy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All women who prepared for abdominal myomectomies will be invited to participate in the study
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
measure will be Mean amount of blood loss | intraoperative
  measure will be Mean amount of blood loss by gravimetric methods

SECONDARY OUTCOMES:
the number of the patients need of blood transfusion | 24 hours post delivery
  calculate the number of the patients need of blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: hany f allam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No